CLINICAL TRIAL: NCT06008899
Title: Efficacy of Ultrasound-assisted Caudal Epidural Pulsed Radiofrequency for Anal and Perineal Pain in Cancer Patients, a Prospective Randomized Clinical Study
Brief Title: Efficacy of Ultrasound-assisted Caudal Epidural Pulsed Radiofrequency for Anal Pain in Cancer Patients,
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Adel El sherif,MD, associate professor of anesthesia, intensive care and pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 629
Record Dates: First submitted 2023-08-17; First posted 2023-08-24 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Perineal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound (US) assisted caudal epidural pulsed radiofrequency (Active Comparator)
  Interventions: Procedure: US assisted caudal epidural pulsed radiofrequency
- conventional medical treatment (No Intervention)

INTERVENTIONS:
Procedure: US assisted caudal epidural pulsed radiofrequency — patients will receive US assisted caudal epidural pulsed radiofrequency and followed up to 8 weeks
  Arms: ultrasound (US) assisted caudal epidural pulsed radiofrequency

SUMMARY:
Our primary goal will be to investigate the analgesic efficacy of ultrasound (US)-assisted caudal epidural PRF (pulsed radiofrequency)( stimulation in patients with perineal or anal pain cancer patients using (visual analog scale (VAS) scores from 0 to 10 at the baseline (pretreatment), two, four, and eight weeks; secondary outcomes will be the effects on opioid use and total opioid use in the 24 h, quality of life, patient satisfaction and opioid and intervention related side effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology physical status of I or III (ASA), of both sex
* cancer-related anal or perineal pain

Exclusion Criteria:

* coagulopathies
* allergies to the contrast dye
* patients with moderate or significant cardiac/respiratory disease or hepatic

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
visual analog scale (VAS) score 4 weeks post-intervention | 8 weeks
  Our primary goal will be to investigate the analgesic efficacy of ultrasound-assisted caudal epidural PRF stimulation in patients with perineal or anal pain cancer patients using VAS scores from 0 to 10 at the baseline (pretreatment), two, four, and eight weeks

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer instIitute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No